CLINICAL TRIAL: NCT06190535
Title: Doses Systematic Per Oral Administration of Etamsylate Can Reduce Postpancreatectomy Hemorrhage From Pancreatic Stump in Pancreatogastrostomy
Brief Title: Can Administration of Etamsylate Reduce Postpancreatectomy Hemorrhage
Acronym: PGPPH1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sfax (Other)
Responsible Party: Principal Investigator, Ali Kchaou, Ali Kchaou MD FACS, University of Sfax
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PGPPH1
Record Dates: First submitted 2023-12-18; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Postpancreatectomy Hemorrhage
MeSH Terms: interventions — Ethamsylate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etamsylate + (Experimental): Arm in which etamsylate (Dicynone injectable 250mg/2ml) is administrated through the nasogastric tube (NT) 2 ampules twice (X2)/day for 48 hours.
  Interventions: Drug: Etamsylate
- the standard postoperative treatment (No Intervention): Arm in which patients have the standard postoperative treatment

INTERVENTIONS:
Drug: Etamsylate — Enteral administration of Etamsylate as solution galenic form
  Arms: Etamsylate +

SUMMARY:
In several studies comparing the tow types of pancreato-digestive anastomosis: pancreatogastrostomy (PG) and pancreatojejunostomy (PJ), authors concluded that PG exposed to more postpancreatectomy hemorrhage (PPH) especially early, digestive and moderate hemorrhage classified as type A according to the classification of the ISGPS.

In this way we try to test the ability of the enteral administration through the nasogastric tube of Etamsylate for 48 hours after Whipple to reduce the rate of digestive PPH and mortality.

DETAILED DESCRIPTION:
Whipple procedure is usually performed for periampullary malignancies. If the mortality of this intervention has been markedly decreased, it persists a morbid one. Morbidity is mainly due to postoperative leak of the pancreato-digestive anastomosis or postoperative pancreatic fistula (POPF), but also to postpancreatectomy hemorrhage (PPH). In several studies comparing the tow types of pancreato-digestive anastomosis: pancreatogastrostomy (PG) and pancreatojejunostomy (PJ), authors concluded that PG exposed to more postpancreatectomy hemorrhage (PPH) especially early, digestive and moderate hemorrhage classified as type A according to the classification of the ISGPS. In this case of hemorrhage, blood generally comes from pancreatic stump which is anastomosed or telescoped in the stomac. Incomplete hemostasis , soft pancreatic tissue and vascular fragility can help PPH to occur.

Etamsylate is an antihemorrhagic agent which works by increasing the resistance in the endothelium of capillaries and stimulating platelet adhesion. It also inhibits synthesis and action of prostaglandins causing platelet disaggregation, vasodilation and increased capillary permeability.

In this way, the investigators try to test the ability of the enteral administration through the nasogastric tube of Etamsylate for 48 hours after Whipple to reduce the rate of digestive PPH and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing Whipple procedure regardless the type of pathology and in which a PG is performed.

Exclusion Criteria:

* Patients undergoing Whipple procedure regardless the type of pathology and in which a PJ is performed.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative early (24-48 hours) digestive hemorrhage | 24-48 hours, postoperative day Day 1, Day 2
  Blood in NT, hematemesis in the postoperative course

SECONDARY OUTCOMES:
Operative mortality | 30 day
  In hospital or 30 day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Kchaou, Sfax, Tunisia

IPD SHARING:
Plan to Share IPD: No